CLINICAL TRIAL: NCT03606213
Title: Safety, Immunogenicty and Anti-Reservoir Activity of an Electroporation-Administered HIV DNA Vaccine Encoding GAG, POL and ENV Proteins With IL-12 Plasmid in HIV-Infected Adults on Antriretroviral Therapy.
Brief Title: Therapeutic Vaccination in Treated HIV Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steven Deeks (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of California, Los Angeles (Other); Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Steven Deeks, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAIDS-ES 38409; U01AI131296 (NIH)
Record Dates: First submitted 2018-07-02; First posted 2018-07-30 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: HIV-1-infection
Keywords: HIV Vaccine; Electroporation
MeSH Terms: interventions — rocakinogene sifuplasmid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A - Arm 1 (Placebo Comparator): Placebo will be administered by electoporation at Day 0 and Weeks 4, 8 and 12
  Interventions: Device: CELLECTRA® 2000
- Cohort A - Arm 2 (Active Comparator): Active gag/pol, env and IL-12 plasmids (PENNVAX-GP and INO-9102)) administered by electoporation (CELLECTRA-2000) at Day 0 and Weeks 4, 8 and 12.
  Interventions: Biological: PENNVAX-GP; Biological: INO-9012; Device: CELLECTRA® 2000
- Cohort A - Arm 3 (Active Comparator): Active gag/pol and IL-12 plasmids (INO-6145 INO-9012) will be administered by electroporation (CELLECTRA-2000) at Day 0 and Weeks 4, 8 and 12.
  Interventions: Biological: INO-6145; Biological: INO-9012; Device: CELLECTRA® 2000
- Cohort B - Arm 1 (Active Comparator): A single arm study of gag/pol/env/IL-12 DNA plasmids PENNVAX-GP and INO-9102) administered by electoporation (CELLECTRA-2000) will be performed in HIV-infected adults for whom ART was initiated during acute HIV infection.
  Interventions: Biological: PENNVAX-GP; Biological: INO-9012; Device: CELLECTRA® 2000

INTERVENTIONS:
Biological: PENNVAX-GP — PENNVAX®-GP is a circular, double stranded, deoxyribonucleic acid consisting of expression plasmids that encode synthetic HIV-1 multiclade consensus Gag, Pol and Env proteins.
  Other Names: HIV DNA vaccine
  Arms: Cohort A - Arm 2; Cohort B - Arm 1
Biological: INO-6145 — INO-6145 is a circular, double stranded, deoxyribonucleic acid consisting of expression plasmids that encode synthetic HIV-1 multiclade consensus Gag and Pol proteins.
  Other Names: HIV DNA vaccine
  Arms: Cohort A - Arm 3
Biological: INO-9012 — The IL-12 DNA adjuvant (INO-9012) consists of a single plasmid containing a dual promoter system for expression of both the IL-12 p35 and p40 genes necessary for production of the active heterodimeric (p70) IL-12 protein.
  Other Names: IL-12 DNA adjuvant
  Arms: Cohort A - Arm 2; Cohort A - Arm 3; Cohort B - Arm 1
Device: CELLECTRA® 2000 — Electroporation (EP) is a technology in which an electrical field is applied to increase the permeability of cell membranes and thereby enhance the uptake of drugs, vaccines, or other agents into target cells. This technology has been used in the last decade in both therapeutics and vaccinations. EP is currently being used to deliver cancer vaccines and therapeutics as well as in gene therapy. The expression levels are increased by as much as 3 orders of magnitude over plasmid injection alone.
  Other Names: Electroporation device

SUMMARY:
The central premise of our program is that durable control of HIV in the absence of antiretroviral therapy ("remission") will require the generation of de novo potent and sustained HIV-specific CD8+ cell responses that target evolutionarily conserved epitopes. Our program is inspired by the recent success of VGX-3100 (Inovio), a DNA therapeutic vaccine for HPV that leads to histopathologic regression of pre-malignant lesions in people and is associated with a potent, sustained boost to HPV-specific CD8+ T cell populations. A closely related multi-clade gag/pol/env DNA vaccine administered with an IL-12 DNA plasmid (PENNVAX, Inovio) has been studied for HIV prevention and is known to be both safe and highly immunogenic. In a randomized placebo-controlled study we will compare the immunogenicity and anti-reservoir activities of gag/pol DNA versus gag/pol/env DNA (both administered with IL-12). We will determine for the first time in established HIV disease whether presence of env in a DNA vaccine blunts T cell responses to more conserved Gag-specific and Pol-specific epitopes. We will also determine if Env-specific responses (which will presumably be mediated by antibodies and antibody-dependent cellular cytotoxicity, or ADCC) have a measurable effect on reservoir.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age ≥ 18 and ≤ 65 years
3. HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen or plasma HIV-1 RNA viral load.
4. For Cohort A participants, ART initiated during chronic infection (e.g., more than 6 months after estimated date of infection, or as determined by site investigator and/or available medical records).
5. For Cohort B participants, ART initiated during "hyperacute" HIV infection (Fiebig I/II) or early HIV infection (Fiebig III/IV).
6. On continuous antiretroviral therapy for at least 24 months without any interruptions of greater than 14 consecutive days, and on a stable regimen for at least 8 weeks, without plans to modify ART during the study period
7. Screening plasma HIV RNA levels < 40 copies/mL on all available determinations in past 24 months (isolated single values ≥ 40 but < 200 copies/mL will be allowed if they were preceded and followed by undetectable viral load determinations)
8. Screening CD4+ T-cell count ≥ 350 cells/mm3
9. Creatinine Clearance (CrCl) > 60 mL/min via Cockroft-Gault method at screening
10. The following laboratory criteria must be met at screening:

    * Absolute neutrophil count (ANC) ≥ 1000 neutrophils/mm3
    * Hemoglobin ≥ 10.0 g/dL
    * Platelet count ≥ 100,000/uL
    * Aspartate aminotransferase (AST) ≤ 2x upper limit of normal (ULN)
    * Alanine aminotransferase (ALT) ≤ 2x ULN

Exclusion Criteria:

1. Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study

a. Acceptable birth control is defined as the following: i. For female participants of childbearing potential, two of the following forms of contraception are required, one of which must be a barrier method:

1. Condoms (male of female) with or without a spermicidal agent 2. Diaphragm or cervical cap with spermicide 3. Intrauterine device (IUD) with published data showing that expected failure rate is < 1% per year 4. Tubal ligation 5. Hormone-based contraceptive such as oral birth control pills ii. Male participants participating in sexual activity that could lead to pregnancy must agree to at least one reliable method of contraception of the above listed 2. Active malignancy requiring systemic chemotherapy or surgery in the preceding 3 months or for whom such therapies are expected in the subsequent 6 months 3. Active (untreated) HCV or HBV infection 4. Decompensated liver disease as defined by the presence of ascites, encephalopathy, esophageal or gastric varices, or persistent jaundice 5. Serious illness requiring systemic treatment and/or hospitalization in the 3 months prior to study enrollment 6. Concurrent treatment with immunomodulatory drugs, and/or exposure to any immunomodulatory drug in the 4 weeks prior to study enrollment (e.g. corticosteroid therapy equal to or exceeding a dose of 15 mg/day of prednisone for more than 10 days, IL-2, interferon-alpha, methotrexate, cancer chemotherapy). NOTE: use of inhaled or nasal steroid is not exclusionary.

7. Serious medical or psychiatric illness that, in the opinion of the site investigator, would interfere with the ability to adhere to study requirements or to give informed consent.

8. Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements or to give informed consent.

9. Unable to undergo leukapheresis procedure 10. Acute or chronic bleeding or clotting disorder that would contraindicate IM injections or use of blood thinners (e.g. anticoagulants or antiplatelet drugs) within 2 weeks of Day 0; 11. Less than two acceptable sites available for IM injection considering the deltoid and anterolateral quadriceps muscles; 12. Tattoos, keloids or hypertrophic scars located within 2 cm of intended treatment site; 13. Cardioverter-defibrillator or pacemaker (to prevent a life-threatening arrhythmia) that is located in ipsilateral deltoid injection site (unless deemed acceptable by a cardiologist); 14. Metal implants or implantable medical device within the intended treatment site (i.e. electroporation area)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deeks, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Zuckerberg San Francisco General Hospital (ZSFG), San Francisco, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort A - Arm 1 | Cohort A - Arm 2 | Cohort A - Arm 3 | Cohort B - Arm 1
Started | 15 | 16 | 14 | 11
Completed | 15 | 16 | 14 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - Arm 1 | Cohort A - Arm 2 | Cohort A - Arm 3 | Cohort B - Arm 1 | Total
Number analyzed (Participants) | 15 | 16 | 14 | 11 | 56
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [44 to 57] | 56 [52 to 60] | 55 [50 to 58] | 44 [34 to 54] | 54 [44 to 57]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex/Gender: Male | 12 | 15 | 13 | 11 | 51
  Sex/Gender: Female | 1 | 0 | 1 | 0 | 2
  Sex/Gender: Non-binary | 1 | 1 | 0 | 0 | 2
  Sex/Gender: Transgender female | 1 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 2 | 3 | 13
  Not Hispanic or Latino | 9 | 11 | 12 | 8 | 40
  Unknown or Not Reported | 0 | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 0 | 2 | 4 | 1 | 7
  White | 7 | 10 | 7 | 8 | 32
  More than one race | 5 | 3 | 2 | 0 | 10
  Unknown or Not Reported | 1 | 1 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 14 | 11 | 56

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Grade 3 or Higher Treatment-related Adverse Events
Description: Counts and percentages of adverse events will be presented in frequency tables and characterized for each arm with 95% Clopper-Pearson Confidence Intervals. We will use the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1
Time Frame: Week 64
Population: All who received at least one dose
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - Arm 1 | Cohort A - Arm 2 | Cohort A - Arm 3 | Cohort B - Arm 1
Number analyzed (Participants) | 15 | 16 | 14 | 11
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: The Change in the Magnitude of T Cell Responses Will be Evaluated by the IFN-γ Enzyme-linked Immunospot (ELISpot) Assay
Description: The magnitude of Gag-specific responses was characterized in detail via matrix mapping using vaccine-matched peptides, while pools of 15 overlapping peptides will used to evaluate the magnitude of T cell response to Pol and Env, as well as Nef (internal control). In addition, ELISpot responses to pools of Gag, Pol, Env, and Nef peptides (n=50 peptides/pool) that have been derived from circulating HIV viruses (potential T cell epitope peptides, PTE; NIH AIDS Reagent Program) were evaluated in parallel. All measures were performed on two baseline PBMC samples. The primary outcome in terms of the magnitude of the response was calculated as the fold-change (ratio) in the number of spot-forming units per million peripheral blood mononuclear cells between week 14 and baseline (pre-vaccine).
Time Frame: Baseline to Week 14
Population: Subjects analyzed by treatment received. Excludes one individual due to poor sample quality at week 14.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Cohort A - Arm 1 | Cohort A - Arm 2 | Cohort A - Arm 3 | Cohort B - Arm 1
Number analyzed (Participants) | 15 | 15 | 12 | 9
Ratio | 0.95 [0.48 to 1.36] | 1.31 [0.94 to 2.07] | 2.37 [1.06 to 3.15] | 1.24 [0.70 to 1.82]
Statistical Analysis 1: Comparison: Cohort A - Arm 1 vs Cohort A - Arm 2 vs Cohort A - Arm 3; Test type: Other; p = 0.56, Wilcoxon (Mann-Whitney) — P-value week 14 versus baseline (Cohort A, arm 1; placebo)

3. Secondary Outcome: HIV Reservoir Size
Description: The frequency of circulating CD4+ T cells harboring replication-competent HIV as measured using multiplex digital droplet PCR assay to quantify the total number of intact proviruses (IPDA). The frequency of cells harboring an intact genome per million CD4+ T cells was calculated. Values were log10 transformed. The mean log10 change from baseline to Week 64 was calculated.
Time Frame: Baseline and Week 64
Measure: Mean (Standard Error); unit: Log10 intact genomes/million CD4 T cells
Arm/Group | Cohort A - Arm 1 | Cohort A - Arm 2 | Cohort A - Arm 3 | Cohort B - Arm 1
Number analyzed (Participants) | 13 | 16 | 10 | 9
Log10 intact genomes/million CD4 T cells | 0.06 (0.08) | -0.09 (0.08) | 0.03 (0.015) | -0.03 (0.01)

ADVERSE EVENTS:
Time Frame: 64 weeks
Description: We conducted structured interviews at each visit
Arm/Group | Cohort A - Arm 1 | Cohort A - Arm 2 | Cohort A - Arm 3 | Cohort B - Arm 1
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/14 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/16 | 2/14 | 1/11
Other Adverse Events (participants affected / at risk) | 15/15 | 16/16 | 14/14 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - Arm 1 (N=15) | Cohort A - Arm 2 (N=16) | Cohort A - Arm 3 (N=14) | Cohort B - Arm 1 (N=11)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidality (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar depression with hypomania (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - Arm 1 (N=15) | Cohort A - Arm 2 (N=16) | Cohort A - Arm 3 (N=14) | Cohort B - Arm 1 (N=11)
Injection site reaction (General disorders) | 15 | 16 | 14 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03606213/Prot_SAP_ICF_001.pdf